CLINICAL TRIAL: NCT00304161
Title: Depression Diagnosis and Treatment in Parkinson Disease
Brief Title: Effectiveness of Antidepressant Treatment for Depression in People With Parkinson's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: K23MH067894 (NIH); K23MH067894 (NIH)
Record Dates: First submitted 2006-03-15; First posted 2006-03-17 (Estimated); Results first posted 2015-03-13 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2016-12

CONDITIONS: Depressive Disorder; Parkinson Disease
Keywords: Depression; Parkinson's Disease; Atomoxetine
MeSH Terms: conditions — Depressive Disorder; Parkinson Disease; Depression | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atomoxetine (Active Comparator): Participants will receive 40-80mgs of atomoxetine orally once daily.
  Interventions: Drug: Atomoxetine
- Placebo (Placebo Comparator): Participants will receive placebo treatment once daily; the pill (taken orally) will resemble the atomoxetine pill but will not contain an active drug.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atomoxetine — 40 to 80 mg orally once daily for 8 weeks
  Other Names: Straterra
  Arms: Atomoxetine
Drug: Placebo — 40 to 80 mg orally once daily for 8 weeks
  Arms: Placebo

SUMMARY:
This study will evaluate the effectiveness of atomoxetine in reducing symptoms of depression in people with Parkinson's disease.

DETAILED DESCRIPTION:
Depression is a serious medical condition that affects people's thoughts, feelings, and ability to function in everyday life. Depression can happen to anyone, but it is more of a risk in people with Parkinson's disease, a progressive brain disorder that is caused by a loss of dopamine-producing brain cells. As many as half of people with Parkinson's may suffer from depression. These individuals experience different symptoms than those who have depression alone. For example, they are prone to higher rates of anxiety, sadness without guilt or self-blame, and lower suicide rates despite high rates of suicidal thoughts. Depression treatment can help people with Parkinson's disease who are depressed to manage both diseases and improve the quality of their lives. This study will evaluate the effectiveness of atomoxetine, an antidepressant medication, in reducing symptoms of depression in people with Parkinson's disease.

Participants in this double-blind study will be randomly assigned to receive either atomoxetine or placebo for 8 weeks. All participants will report to the study site at baseline and Weeks 2, 4, and 8. Psychiatric, neuropsychological, and neurological assessments will be performed, including evaluations with the Inventory of Depressive Symptomatology (IDS) scale and the Clinical Global Impression-Improvement (CGI-I) scale. All participants will be offered continued routine psychiatric care with the study physician upon completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson's disease
* IDS score greater than 21
* Mini-Mental State Examination (MMSE) score greater than 15

Exclusion Criteria:

* Recent deep brain stimulation
* Currently participating in an antidepressant trial at a less than adequate dose and duration
* Severe depression or depression with suicide ideation
* History of liver toxicity
* Unstable medical disease or comorbid psychiatric disease

Ages: 30 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2004-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Weintraub, MD, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - Philadelphia Veterans Affairs Medical Center, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Weintraub D, Mavandadi S, Mamikonyan E, Siderowf AD, Duda JE, Hurtig HI, Colcher A, Horn SS, Nazem S, Ten Have TR, Stern MB. Atomoxetine for depression and other neuropsychiatric symptoms in Parkinson disease. Neurology. 2010 Aug 3;75(5):448-55. doi: 10.1212/WNL.0b013e3181ebdd79. PMID 20679638
- See also: Manuscript — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC2918470/pdf/7887.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from The Parkinson's Disease and Movement Disorders Center at Pennsylvania Hospital and the Parkinson's Disease Research, Education, and Clinical Center at the Philadelphia Veterans Affairs Medical Center between 2004-2009.
Period: Overall Study
Arm/Group | Atomoxetine | Placebo
Started | 28 | 27
Completed | 22 | 21
Not Completed | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Atomoxetine: Participants will receive atomoxetine treatment
- Placebo: Participants will receive placebo treatment
- Total: Total of all reporting groups
Arm/Group | Atomoxetine | Placebo | Total
Number analyzed (Participants) | 28 | 27 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 11 | 25
  >=65 years | 14 | 16 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (9.5) | 64.9 (11.5) | 64.3 (10.5)
Gender [Count of Participants; unit: Participants]
  Female | 8 | 11 | 19
  Male | 20 | 16 | 36
Region of Enrollment [Number; unit: participants]
  United States | 28 | 27 | 55

OUTCOME MEASURES:

1. Primary Outcome: Inventory of Depressive Symptomatology- Clinician Rated (IDS-C) Scale
Description: The primary measure of depression symptom severity was the Inventory for Depressive Symptomatology-Clinician Rated (IDS-C), a 30-item (scores 0-84, increasing scores indicating greater depression severity) comprehensive instrument that is increasingly used as a primary outcome measure in major depression treatment studies in the general population. An IDS-C score of greater than or equal to 22 was indicative of at least moderate depression. The IDS-C was administered at every study visit. The criteria for the primary measure of treatment response was a >50% decrease in IDS-C score from baseline.
Time Frame: Week 8
Measure: Number; unit: percentage of improved participants
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 22 | 21
percentage of improved participants | 22.7 | 9.5

2. Secondary Outcome: Clinical Global Impression-Improvement Scale
Description: The Clinical Global Impression-Improvement scale rates total improvement on a 7 point scale:
  1. = Very much improved
  2. = Much improved
  3. = Minimally improved
  4. = No change
  5. = Minimally worse
  6. = Much worse
  7. = Very much worse
  A participant scoring a 1 or 2 is considered a responder on the CGI scale.
Time Frame: Week 8
Measure: Number; unit: percentage of responders
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 22 | 21
percentage of responders | 45.5 | 33.3

ADVERSE EVENTS:
Arm/Group | Atomoxetine | Placebo
Serious Adverse Events (participants affected / at risk) | 2/28 | 2/27
Other Adverse Events (participants affected / at risk) | 7/28 | 6/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Atomoxetine (N=28) | Placebo (N=27)
Suicide Ideation (Psychiatric disorders) | 1 | 0
Congestive Heart Failure (Cardiac disorders) | 1 | 0
Chest Pain (Cardiac disorders) | 0 | 1
Urosepsis (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Atomoxetine (N=28) | Placebo (N=27)
Constipation (Gastrointestinal disorders) | 7 | 1
Nausea/Vomiting (Gastrointestinal disorders) | 0 | 5

LIMITATIONS AND CAVEATS:
First, the sample size was relatively small. Second, the diagnostic criteria for depression which are typically used in clinical trials were not used as an inclusion criterion. Third, antidepressant use at baseline was common in our population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No